CLINICAL TRIAL: NCT01198171
Title: The Relationship of Racial Genetic Admixture With Endometrial Cancer Outcomes
Brief Title: Racial and Genetic Biomarkers of Response in Tissue Samples From Patients With Endometrial Cancer
Status: Completed | Type: Observational
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: GOG Foundation (Network)
Other Study IDs: GOG-8022; NCI-2011-02867 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000684547; GOG-8022; GOG-8022 (Other: Gynecologic Oncology Group); GOG-8022 (Other: CTEP); P50CA134254 (NIH); R01CA071754 (NIH); R21CA133295 (NIH); U10CA027469 (NIH); U10CA037517 (NIH)
Record Dates: First submitted 2010-09-08; First posted 2010-09-09 (Estimated); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Stage I Uterine Corpus Cancer; Stage II Uterine Corpus Cancer; Stage III Uterine Corpus Cancer; Stage IV Uterine Corpus Cancer

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Basic science (DNA analysis): DNA from archived frozen normal tissue samples is genotyped for the ancestry informative markers. Clinicopathological and demographic characteristics associated with each sample are also collected.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Study of Socioeconomic and Demographic Variables

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Study of Socioeconomic and Demographic Variables

SUMMARY:
This research study is studying racial and genetic biomarkers of response in tissue samples from patients with endometrial cancer. Studying samples of tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer. DNA analysis of tumor tissue may also help doctors predict how well patients will respond to treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To identify racial categorization as the proportion of genetic background of African-American or European-American women with endometrioid endometrial cancer (EEC).

II. To evaluate the association of racial genetic admixture with clinicopathologic variables and outcomes.

SECONDARY OBJECTIVES:

I. To compare the concordance between racial genetic admixture and self-designated race categorization.

OUTLINE: This is a multicenter study. Patients are stratified by race (African-American vs European-American) and disease stage (I vs II vs III vs IV).

DNA from archived frozen normal tissue samples is genotyped for the ancestry informative markers. Clinicopathological and demographic characteristics associated with each sample are also collected.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed endometrial cancer

  * Stage I-IV disease regardless of grade
  * Underwent surgical staging including hysterectomy, bilateral oophorectomy, washings, and pelvic lymphadenectomy
* Eligible and evaluated on GOG-0210 clinical trial, a Molecular Staging Study in Endometrial Cancer
* Available frozen or formalin-fixed and paraffin-embedded normal tissue that is free of tumor cells and yields sufficient high-quality normal DNA for testing
* Consented their specimens and clinical data to be collected and used in future studies
* Self-declared African-American or Caucasian race

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient with endometrial cancer
Sampling Method: Non-Probability Sample
Enrollment: 243 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Clinicopathologic and demographic characteristics: characteristics: self-reported race, stage, age, race, parity, body-mass index, stage, grade, depth of invasion, lymph-vascular space invasion, and metastasis | 1 year
Overall survival | 1 year
Progression-free survival | 1 year
Proportion of genetic background that is of African-American descent | 1 year

SECONDARY OUTCOMES:
Racial genetic admixture score, summarized by race and other clinicopathologic variables | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Rodney Rocconi, Principal Investigator — Gynecologic Oncology Group
Locations (1):
- Gynecologic Oncology Group, Philadelphia, Pennsylvania, United States